CLINICAL TRIAL: NCT01541670
Title: A Study to Assess the Safety and Tolerability of Anti-MIF Antibody in Subjects With Lupus Nephritis
Brief Title: Safety Study of Anti-Macrophage Migration Inhibitory Factor (Anti-MIF) Antibody in Lupus Nephritis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 391001
Record Dates: First submitted 2012-02-20; First posted 2012-03-01 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-label Dose-Escalation Arm (Experimental): Conducted in an ascending dose manner, subjects will be assigned to single- or multiple-dose administration of the investigational product
  Interventions: Drug: Anti-Macrophage Migration Inhibitory Factor (Anti-MIF) Antibody

INTERVENTIONS:
Drug: Anti-Macrophage Migration Inhibitory Factor (Anti-MIF) Antibody — Intravenous injection

SUMMARY:
The purpose of this study is to determine the safety and tolerability of Anti-MIF Antibody in subjects with lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent obtained from the subject
* Males and females of age 18 years and older at the time of screening
* Established diagnosis of systemic lupus erythematosus (SLE) according to the American College of Rheumatology classification criteria
* Documented renal biopsy evidence of proliferative glomerulonephritis prior to screening
* Urine protein-to-creatinine ratio > 0.5 (mg/mg)

Exclusion Criteria:

* Any significant health problem other than lupus or lupus nephritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-11-28 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing serious adverse events (SAEs) and/or adverse events (AEs) regardless of causality | Week 21

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters | Week 21
  Maximum concentration (Cmax), minimum concentration (Cmin), area under the curve (AUC), half-life (t1/2), clearance (CL) , mean residence time (MRT), volume of distribution at steady state (Vdss)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (23):
- United States (11):
  - Academic Medical Research Institute Inc., Los Angeles, California
  - Mohamed A. El-Shahawy, Los Angeles, California
  - North Valley Nephrology, Yuba City, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - University of Colorado, Denver, Colorado
  - Tulane University Hospital & Clinic, New Orleans, Louisiana
  - Clinical Research Development Associates, LLC, Springfield Gardens, New York
  - Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Ramesh Gupta, Memphis, Tennessee
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
- Australia (3):
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Canada (2):
  - CHUM Hôpital Saint-Luc, Montreal, Quebec
  - St. Paul´s Hospital, Saskatoon, Saskatchewan
- Mexico (5):
  - Mexico Center for Clinical Research S.A de C.V, Mexico City, Mexico City
  - Hospital y Clinica OCA SA de CV, Monterrey, Nuevo León
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Clinica San Jose, Sonora, Obregon
  - Hospital CIMA Chihuahua, Chihuahua City
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland